CLINICAL TRIAL: NCT00951002
Title: A Multicenter Clinical Trial to Evaluate the Efficacy of Human Acellular Dermal Matrix in the Treatment of Anal Fistula
Brief Title: The Efficacy of Human Acellular Dermal Matrix in the Treatment of Anal Fistula
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhen Jun Wang (Other)
Collaborators: Second Affiliated Hospital of Medical College Shandong University (Other); Beijing Anorectal Hospital (Other); The Central Hospital of China Aerospace Corporation (Unknown); Children's Hospital of Hebei Province (Other); The 85th Hosptial of P.L.A (Unknown); Shandong Provincial Hospital (Other Government); Peking University Third Hospital (Other); Shenzhen People's Hospital (Other); The Second Artillery General Hospital (Other); Dongzhimen Hospital, Beijing (Other); Shenyang Anorectal Hospital (Other); Wuhan Iron and Steel Workers' Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhen Jun Wang, Professor and Chief of General Surgery, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Other Study IDs: AF-HADM-01
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Anal Fistula; Treatment; Postoperative Complications; Acellular Dermal Matrix
Keywords: anal fistula; acellular dermal matrix; treatment; postoperative complications; recurrence
MeSH Terms: conditions — Rectal Fistula; Postoperative Complications; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acellualr dermal matrix: patients treated with acellular dermal matrix plug
  Interventions: Procedure: acellular dermal matrix plug

INTERVENTIONS:
Procedure: acellular dermal matrix plug — anal fistula treated with human acellular dermal matrix plug
  Other Names: Ruinuo

SUMMARY:
The purpose of this study is to determine whether human acellular dermal matrix plug is effective in the treatment of anal fistula

DETAILED DESCRIPTION:
Recently, the use of biomaterial for the treatment of anal fistula has drawn great interest. The advantages of this technique include simple and repeatable application, preservation of sphincter integrity, minimal patient discomfort, and the ability for subsequent surgical options if needed. Champagne et al reported using a biologic absorbable anal fistula plug which is made from lyophilized porcine small intestinal submucosa (Surgisis®). In their series of 46 patients treated with the anal fistula plug, a success rate of 83 percent was achieved at a median follow-up of 12 months. In addition, evaluation of the functional outcome after fistula closure showed no impairment of continence with significant improvement in quality of life showed. However, the long term success rates of Surgisis® are variable according to other studies.

Human acellular dermal matrix (ADM) is a biologic material consists of dermis without its cellular components. Early and rapid revascularization of the implanted ADM, as was shown in our previous experimental study, is thought to enhance resistance to infection and contamination. These properties make ADM an attractive alternative for the treatment of anal fistula. The ability of ADM to become vascularized and remodeled by autologous cells may be advantageous for anal fistulas healing.

The purpose of this study is to determine whether human acellular dermal matrix plug is effective in the treatment of anal fistula.

ELIGIBILITY:
Inclusion Criteria:

* complex anal fistula

Exclusion Criteria:

* pregnancy or lactation
* with operation contraindication
* allergic constitution to heterogeneous protein
* complicated with tumor
* complicated with acute infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients with complex anal fistula
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 01/07/2011

SECONDARY OUTCOMES:
recurrence rate | 01/07/2011

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Jun Wang, M.D., Study Chair — Beijing Chao Yang Hospital; Ke Ding, M.D., Principal Investigator — Second Affiliated Hospital of Medical College Shandong University; Chang Shun Wang, M.D., Principal Investigator — Beijing Anorectal Hospital; Li Yong Wang, M.D., Principal Investigator — The Central Hospital of China Aerospace Corporation; Li Ya Wang, M.D., Principal Investigator — Children's Hospital of Hebei Province; Min Kong, M.D., Principal Investigator — The 85th Hosptial of P.L.A; Xue Zhi Xin, M.D., Principal Investigator — Shandong Provincial Hospital; Chao Wen Chen, M.D., Principal Investigator — Peking University Third Hospital; Xiao Dong Yang, M.D., Principal Investigator — Shenzhen People's Hospital; Ke Zhao, M.D., Principal Investigator — The Second Artillery General Hospital; Bao Ming Zhao, M.D., Principal Investigator — Dongzhimen Hospital, Beijing; Xian Dong Zeng, M.D., Principal Investigator — Shenyang Anorectal Hospital; Si Tu Guang Wei, M.D., Principal Investigator — Wuhan Iron and Steel Workers' Hospital
Locations (13):
- China (13):
  - Beijing Anorectal Hospital, Beijing, Beijing Municipality
  - Dongzhimen Hospital Affiliated to Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Central Hospital of China Aerospace Corporation, Beijing, Beijing Municipality
  - The Second Artillery General Hospital, Beijing, Beijing Municipality
  - General Surgery, Beijing Chao Yang Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Hebei Children's Hospital, Shijiazhuang, Hebei
  - General Staff Hospital of Wuhan Iron and Steel (Group) Corp, Wuhan, Hubei
  - Shenyang Anorectal Hospital, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Second Affiliated Hospital of Medical College Shandong University, Jinan, Shandong
  - The 85th Hosptial of P.L.A, Shanghai, Shanghai Municipality

REFERENCES:
- [Background] Han JG, Xu HM, Song WL, Jin ML, Gao JS, Wang ZJ, Yang XQ. Histologic analysis of acellular dermal matrix in the treatment of anal fistula in an animal model. J Am Coll Surg. 2009 Jun;208(6):1099-106. doi: 10.1016/j.jamcollsurg.2009.02.052. Epub 2009 Apr 24. PMID 19476898
- [Result] Song WL, Wang ZJ, Zheng Y, Yang XQ, Peng YP. An anorectal fistula treatment with acellular extracellular matrix: a new technique. World J Gastroenterol. 2008 Aug 14;14(30):4791-4. doi: 10.3748/wjg.14.4791. PMID 18720541